CLINICAL TRIAL: NCT02725918
Title: Randomized Phase II Study of Pemetrexed Alone vs Pemetrexed Plus Cisplatin in Patients With EGFR Mutation-positive Advanced NSCLC After First Line EGFR-TKIs Failure
Brief Title: Pemetrexed vs Pemetrexed Plus Cisplatin in EGFR-mutant NSCLC Patients After First Line EGFR-TKIs Failure
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Association of Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTONG1510
Record Dates: First submitted 2016-03-11; First posted 2016-04-01 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC; EGFR-TKI failure; chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Cisplatin

ARMS (2):
- Pem mono (Experimental): Patients in arm B will receive pemetrexed (500 mg/m2, d1) every 3 weeks until PD or intolerable toxicities.
  Interventions: Drug: Pemetrexed
- Pem+Cis (Active Comparator): Patients in arm A will receive 4 cycles of cisplatin (75 mg/m2, d1) and pemetrexed (500 mg/m2, d1) every 3 weeks, those without disease progression (PD) and being tolerable judged by investigator will continue single-agent pemetrexed (500 mg/m2, d1) every 3 weeks as maintenance until progression or intolerable toxicities.
  Interventions: Drug: Pemetrexed; Drug: Cisplatin

INTERVENTIONS:
Drug: Pemetrexed — 500 mg/m2,iv,d1,q3w,until PD
  Other Names: Alimta，pemetrexed disodium
Drug: Cisplatin — 75 mg/m2,iv,d1,q3w,×4 cycles
  Other Names: DDP，platinol
  Arms: Pem+Cis

SUMMARY:
The study is a prospective, multi-center, open-label, randomized, and controlled phase II clinical trial. The investigators hope to figure out the better chemotherapy regimen for the post-EGFR-TKI failure setting. The primary objective of this trial is to compare progression-free survival without grade 4 (G4PFS) toxicities between pemetrexed-cisplatin and single-agent pemetrexed treatment arms.

The trial will include stage IIIB/IV EGFR mutation positive NSCLC patients who got disease progression after front-line EGFR TKI treatment.Eligible patients will be randomized to 2 arms. Patients in arm A will receive 4 cycles of cisplatin (75 mg/m2, d1) and pemetrexed (500 mg/m2, d1) every 3 weeks, those without disease progression (PD) and being tolerable judged by investigator will continue single-agent pemetrexed (500 mg/m2, d1) every 3 weeks as maintenance until progression or intolerable toxicities. Patients in arm B will receive pemetrexed (500 mg/m2, d1) every 3 weeks until PD or intolerable toxicities.

DETAILED DESCRIPTION:
The study is a prospective, multi-center, open-label, randomized, and controlled phase II clinical trial.

The trial will include stage IIIB/IV EGFR activating mutation positive NSCLC patients who got disease progression after frontline EGFR-TKI treatment. Clinical staging is determined according to the routine protocol, which includes enhanced chest CT scans, abdominal ultrasonography or CT scans, brain MRI or CT, and bone scintigraphy. Positron emission tomography (PET)/CT scan is optional. Measurement of acquired resistance to EGFR-TKIs is based on Jackman criteria.

Eligible patients will be randomized to 2 arms. Patients in arm A will receive 4 cycles of cisplatin (75 mg/m2, d1) and pemetrexed (500 mg/m2, d1) every 3 weeks, those without disease progression (PD) and being tolerable judged by investigator will continue single-agent pemetrexed (500 mg/m2, d1) every 3 weeks as maintenance until progression or intolerable toxicities. Patients in arm B will receive pemetrexed (500 mg/m2, d1) every 3 weeks until PD or intolerable toxicities. All patients will be administrated with vitamin B12 and folic acid supplement (vitamin B12 1mg intramuscular injection at least 7 days prior to the first dose of pemetrexed and repeated approximately every 9 weeks during pemetrexed treatment till 22 days after the last dose of pemetrexed; folic acid 0.5 mg orally administered once daily from at least 7 days prior to the first dose of pemetrexed till 22 days after the last dose of pemetrexed).

Efficacy data will be analyzed by intention-to-treat (ITT) population using all randomized patients, and safety data will be evaluated using CTCAE v4.0 criteria for patients who received ≥ 1 dose of study treatment. If the criteria for drug administration (absolute neutrophil count ≥1500/μl, platelets ≥100 000/μl, creatinine clearance ≥45 ml/min, no grade ≥3 nonhematologic toxicity [except for alopecia]) were not met, drug administration have to be delayed to allow sufficient time for recovery. If a delay of more than 42 days due to toxicity was necessary, the patient will be discontinued from the study. Dose adjustments according to hematologic toxicity at the start of a subsequent cycle of the therapy will be based on platelet and neutrophil nadir counts from the preceding cycle. Granulocyte colony-stimulating factor is allowed to use for neutropenia event. Patients will be discontinued from study treatment for the following reasons: disease progression; unacceptable toxicities; patient's refusal to continue.

Radiological examinations (according to the RECIST 1.1 criteria) at baseline will be repeated for tumor response evaluation following every two cycles of chemotherapy. Patients will be followed up to 30 days after the last dose of study chemotherapy, and then every 3 months.

Blood samples [8ml with ehylene diamine tetraacetic acid (EDTA) as anticoagulant each time] will be collected at the time of baseline, tumor response evaluation every 2 cycles, and disease progression. Blood samples at baseline and disease progression are mandatory to be provided. Tumor samples collection at the time of baseline and/or disease progression is strongly recommended but not mandatory for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent must be signed.
2. Age of ≥18 and < 75 years old.
3. Performance status (PS) 0 - 2 on the Eastern Cooperative Oncology Group (ECOG) Scale.
4. Histologically confirmed stage IIIB/IV advanced NSCLC harboring activating EGFR mutation.
5. Chemotherapy-naïve for advanced disease.
6. Acquired resistance is measured according to the Jackman criteria. Achieved complete remission (CR)/partial remission (PR)≥4 months or stable disease (SD)>6 months with first-line EGFR TKIs (Gefitinib or Erlotinib or Icotinib) for advanced NSCLC.
7. Disease progression(RECIST) <4 weeks prior to study randomization.
8. Adequate organ function including the following:

   * Bone marrow: absolute neutrophil count (ANC) ≥1.5 x 109/L, platelets ≥100 x 109/L hemoglobin ≥9 g/dL.
   * Hepatic: total bilirubin ≤1.5 times the upper limit of normal (ULN), liver transaminases: aspartate transaminase (AST or SGOT) and alanine transaminase (ALT or SGPT) ≤2.5 times ULN. AST and ALT ≤ 5 x ULN may be included only if Patient has liver metastasis.
   * Renal: calculated creatinine clearance ≥45 mL/min (using the standard Cockcroft-Gault formula).
9. Patients have resolution to <Grade 2 by the CTCAE (Version 4.0), of all clinically significant toxic effects of prior anti-cancer therapy (with the exception of rash and alopecia).
10. Patients with stable central nervous system (CNS) metastasis successfully treated with local therapy, or with asymptomatic CNS metastasis are eligible. Treated stable CNS metastases are allowed; the patient must be stable after radiotherapy for ≥2 weeks and off of corticosteroids for ≥1 week.
11. At least one measurable lesion as defined by RECIST 1.1 criteria.
12. Previous palliative radiation therapy is allowed, but limited in <25% of the bone marrow and must not have included whole pelvis radiation. Patients must have recovered from the toxic effects of the treatment prior to study enrollment (except for alopecia). Prior radiotherapy must be completed one month before study entry. Radiotherapy should not be administered to target lesions selected for this study, unless progression of the selected target lesions within the radiation portal is documented.
13. Estimated life expectancy of at least 8 weeks.
14. For women: must be surgically sterile, postmenopausal, or compliant with a highly effective contraceptive method during and for 3 months after the treatment period; must not be pregnant and must not be lactating; negative pregnancy test is required for women of childbearing potential. Postmenopausal women must have been amenorrhoeic for at least 12 months to be considered of non-childbearing potential. For men: must be surgically sterile or compliant with a highly effective contraceptive method during and for 3 months after the treatment period.
15. Patient compliance and geographic proximity that allow adequate follow-up. Willingness to provide blood samples for EGFR mutation test at baseline and disease progression.

Exclusion Criteria:

1. Patient got disease relapsed within 12 months after post-operative adjuvant chemotherapy, thereafter got failure from subsequent EGFR-TKI treatment cannot be enrolled.
2. History of another malignancy within the last 5 years except cured carcinoma in-situ of uterine cervix, cured basal cell carcinoma of skin and superficial bladder tumors [Ta, Tis & T1].
3. Any unstable systemic disease (including active infection, hepatic, renal or metabolic disease) or serious concomitant disorders that will compromise the safety of the patient, or compromise the patient's ability to complete the study, at the discretion of the investigator.
4. Significant cardiovascular event: congestive heart failure >New York Heart Association (NYHA) class 2; unstable angina, active coronary artery disease (myocardial infarction more than 1 year prior to study entry is allowed); serious cardiac arrhythmia requiring anti-arrythmic therapy ( beta blockers or digoxin are permitted) or uncontrolled hypertension.
5. History of significant neurological or mental disorder, including seizures or dementia.
6. Incision from operation has not healed before the start of study treatment (Small incision for biopsy is eligible.)
7. Presence of clinically uncontrollable third-space fluid collections, for example, ascites or pleural effusions that cannot be controlled by drainage or other procedures prior to study entry.
8. Inability or unwillingness to interrupt aspirin or other non-steroidal anti-inflammatory drugs (NSAIDs) from 2 days before to 2 days after administration of pemetrexed. If a patient is taking an NSAID (including Cox-2 inhibitors) or salicylate with a long half-life (e.g. naproxen, piroxicam, diflusinal, nabumetone, rofecoxib, or celecoxib), it should not be taken from 5 days before to 2 days after the administration of pemetrexed.
9. Inability or unwillingness to take folic acid, vitamin B12 supplementation, or dexamethasone.
10. Inability to comply with protocol or study procedures.
11. Concurrent use of any other anti-tumor therapy during study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-04-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival without grade 4 (G4PFS) | From the date of randomization to the earliest occurrence of the first of grade 4 adverse events (AEs), disease progression, or death from any cause, regardless of whether or not the event leads to discontinuation,assessed up to 4 months.

SECONDARY OUTCOMES:
Progression free survival (PFS) | From the date of randomization to the first date of documented objective progression disease or of death from any cause,assessed up to 6 months.
Overall survival (OS) | From the date of randomization to the date of death from any cause,assessed up to 12 months.
Overall response rate (ORR) | From randomization to date of objective disease progression,assessed up to 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Yi long Wu, Principal Investigator — Guangzhou lung cancer institute
Locations (1):
- Guangdong Lung cancer institute, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zeng Z, Yan HH, Zhang XC, Zhong WZ, He YY, Guan JL, Niu FY, Xie Z, Huang YS, Xu CR, Dong S, Wu YL. Reduced chemotherapy sensitivity in EGFR-mutant lung cancer patient with frontline EGFR tyrosine kinase inhibitor. Lung Cancer. 2014 Nov;86(2):219-24. doi: 10.1016/j.lungcan.2014.09.008. Epub 2014 Sep 18. PMID 25263853
- [Result] Tseng JS, Yang TY, Chen KC, Hsu KH, Yu CJ, Liao WY, Tsai CR, Tsai MH, Yu SL, Su KY, Chen JJ, Chen HY, Chang GC. Prior EGFR tyrosine-kinase inhibitor therapy did not influence the efficacy of subsequent pemetrexed plus platinum in advanced chemonaive patients with EGFR-mutant lung adenocarcinoma. Onco Targets Ther. 2014 May 23;7:799-805. doi: 10.2147/OTT.S62639. eCollection 2014. PMID 24920920
- [Result] Yang JJ, Chen HJ, Yan HH, Zhang XC, Zhou Q, Su J, Wang Z, Xu CR, Huang YS, Wang BC, Yang XN, Zhong WZ, Nie Q, Liao RQ, Jiang BY, Dong S, Wu YL. Clinical modes of EGFR tyrosine kinase inhibitor failure and subsequent management in advanced non-small cell lung cancer. Lung Cancer. 2013 Jan;79(1):33-9. doi: 10.1016/j.lungcan.2012.09.016. Epub 2012 Oct 15. PMID 23079155
- [Result] Zinner RG, Obasaju CK, Spigel DR, Weaver RW, Beck JT, Waterhouse DM, Modiano MR, Hrinczenko B, Nikolinakos PG, Liu J, Koustenis AG, Winfree KB, Melemed SA, Guba SC, Ortuzar WI, Desaiah D, Treat JA, Govindan R, Ross HJ. PRONOUNCE: randomized, open-label, phase III study of first-line pemetrexed + carboplatin followed by maintenance pemetrexed versus paclitaxel + carboplatin + bevacizumab followed by maintenance bevacizumab in patients ith advanced nonsquamous non-small-cell lung cancer. J Thorac Oncol. 2015 Jan;10(1):134-42. doi: 10.1097/JTO.0000000000000366. PMID 25371077